CLINICAL TRIAL: NCT01617369
Title: A Study to Characterize the Durability of Hypertonic Saline for the Enhancement of Mucociliary Clearance in Healthy Subjects
Brief Title: Study to Characterize the Durability of Hypertonic Saline to Enhance Mucociliary Clearance in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Scott Donaldson, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11-1932
Record Dates: First submitted 2012-06-06; First posted 2012-06-12 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2014-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Subjects completed mucociliary clearance measurements (via gamma scintigraphy) at baseline, 30 minutes after inhaling 2.8% NaCl, and 4 hours after inhaling 2.8% NaCl at separate study visits to characterize acute vs. sustained effects of inhaled 2.8% NaCl on this physiologic process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Acute Hypertonic Saline Effect (Experimental): 2.8% NaCl inhaled 30 minutes before Mucociliary Clearance measured.
  Interventions: Device: Hypertonic Saline
- Sustained Hypertonic Saline Effect (Active Comparator): 2.8% NaCl inhaled 4 hours before Mucociliary Clearance measured.
  Interventions: Device: Hypertonic Saline

INTERVENTIONS:
Device: Hypertonic Saline — 2.8% NaCl x 4ml via nebulizer

SUMMARY:
The purpose of this research study is to learn about how long hypertonic saline (HS) works in healthy subjects. Inhaled hypertonic saline is one of the medications used to treat Cystic Fibrosis (CF). In CF and more common lung diseases like chronic bronchitis, mucus builds up in the lungs. Hypertonic saline and other medications currently being developed may help patients with these lung diseases by speeding up mucus clearance from the lung. For these treatments to be effective, they likely need to be able to act for at lease several hours. Investigators are able to measure how lung treatments like hypertonic saline work by conducting a Mucociliary Clearance (MCC) scan. Currently, the investigators do not know how long hypertonic saline works in people who do not have CF. Investigators plan to use this information to improve the design and testing of new treatments for patients with chronic bronchitis.

Objectives:

1. The investigators will use MCC measurements to determine the durability of action of hypertonic saline in healthy (i.e. non-CF) subjects.
2. The investigators will determine the intra- and inter-individual variability of baseline MCC measurements using a slow inhalation/large particle protocol in healthy subjects to guide future sample size calculations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, without respiratory or cardiac comorbidities
* Age 18-55 years, inclusive
* FEV1 > 80% predicted and FEV1/FVC ratio >70%
* Non-pregnant female subjects must be either not sexually active, post-menopausal, surgically sterilized, or agree to use an appropriate "double-barrier" method (such as a diaphragm and condom); or, must currently be using a prescribed transdermal, injection, implant, or oral contraceptive during study participation
* Subjects who are capable of providing their written informed consent to participate in the study

Exclusion Criteria:

* History of smoking > 10 pack-years
* Any history of smoking within 60 days of screening
* Acute upper or lower respiratory illness within 30 days of screening
* Respiratory medication for any indication within 30 days of screening
* History of asthma, chronic bronchitis, or other chronic lung disease
* History of intolerance to hypertonic saline
* Women who are pregnant, lactating, or of childbearing potential who are unwilling to use an acceptable method of contraception throughout the duration of the study.
* Any condition that, in the opinion of the investigator, would potentially jeopardize the safety of the participant or the integrity of the study
* History of radiation exposure within the past year that would cause the subject to exceed limits for adults established by Federal Regulations
* Subjects who, in the opinion of the Principal Investigator, should not participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Donaldson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypertonic Saline: 2.8% NaCl
  Hypertonic Saline: 2.8% NaCl x 4ml via nebulizer
Period: Overall Study
Arm/Group | Hypertonic Saline
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy subjects of any ethnicity between 18-55 years of age, without respiratory or cardiac comorbidities, FEV1 greater than or equal to 80% predicted, FEV1/FVC ratio greater than 70%, non-pregnant female subjects, and subjects who are capable of providing their written informed consent.
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 31.5 [20 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 7
  East Asian | 0
  Black/African American | 3
  West Asian | 0
  Hispanic | 2
  Other, Specify | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Current Smoker [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Whole Lung Mucociliary Clearance
Description: The primary outcome of mucociliary clearance (MCC) will be depicted by calculating the average rate of isotope clearance (%) from the whole lung compartment, measured for 90 minutes after isotope inhalation (MCC-Ave 90), using data points collected every 10 minutes.
  Absolute change in MCC-Ave90 from baseline reported for each arm
Time Frame: 30 minutes and 4 hours after inhalation
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: % Clearance
Groups:
- Acute Hypertonic Saline Effect: 2.8% NaCl inhaled 30 minutes before MCC scan performed
  Hypertonic Saline: 2.8% NaCl x 4ml via Pari LC STAR jet nebulizer
- Sustained Hypertonic Saline Effect: 2.8% NaCl Inhaled 4 hours before mucociliary clearance measured
  Hypertonic saline = 2.8% NaCl x 4 ml delivered via Pari LC STAR jet nebulizer
Arm/Group | Acute Hypertonic Saline Effect | Sustained Hypertonic Saline Effect
Number analyzed (Participants) | 12 | 12
% Clearance | 0.6 (6.4) | -4.0 (5.5)
Statistical Analysis 1: Comparison: Acute Hypertonic Saline Effect vs Sustained Hypertonic Saline Effect; Paired t-test performed. Null hypothesis is that no difference in clearance 30 min and 4 hr after HS inhalation exists; Test type: Superiority; p < .05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Acute Hypertonic Saline Effect | Sustained Hypertonic Saline Effect
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less